CLINICAL TRIAL: NCT00005635
Title: A Phase II Trial to Investigate the Pharmacokinetics, Safety, and Tolerability of Herceptin Administered Subcutaneously in Combination With Paclitaxel in Women With HER2 Overexpressing Metastatic Breast Cancer
Brief Title: Trastuzumab Plus Paclitaxel in Treating Women With Metastatic Breast Cancer That Overexpresses HER2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000067790; MSKCC-99118; GENENTECH-H1994g; NCI-G00-1769
Record Dates: First submitted 2000-05-02; First posted 2004-03-16 (Estimated); Last update posted 2013-08-20 (Estimated); Status verified 2013-08

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; Paclitaxel

INTERVENTIONS:
Biological: trastuzumab
Drug: paclitaxel

SUMMARY:
RATIONALE: Monoclonal antibodies, such as trastuzumab, can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining monoclonal antibody therapy with chemotherapy may kill more tumor cells.

PURPOSE: Randomized phase II trial to study the effectiveness of two different regimens of trastuzumab plus paclitaxel in treating women who have metastatic breast cancer that overexpresses HER2.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the safety and tolerability of subcutaneous trastuzumab (Herceptin) plus paclitaxel in women with HER2 overexpressing metastatic breast cancer. II. Assess the activity of this treatment regimen in these patients. III. Determine the pharmacokinetics of trastuzumab and paclitaxel in this regimen.

OUTLINE: This is a randomized, open label, multicenter study. Patients are randomized to one of two treatment arms. Patients receive a loading dose of trastuzumab (Herceptin) IV over 90 minutes followed by paclitaxel IV over 3 hours on day 0. Paclitaxel is repeated every 3 weeks for 6 courses in the absence of disease progression or unacceptable toxicity. Arm I: Patients receive trastuzumab subcutaneously (SC) weekly starting day 7. Arm II: Patients receive trastuzumab SC twice weekly starting day 7. Treatment with trastuzumab SC continues for 48 weeks in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 80 patients (40 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: HER2 overexpressing (3+) metastatic breast cancer by immunohistochemistry, or amplified by fluorescent in situ hybridization (FISH) No prior chemotherapy for breast cancer metastases No bilateral disease Bidimensionally measurable disease At least 1 target lesion greater than 1 cm2 No significant lymphedema in the arm ipsilateral to mastectomy site, unless patient has an indwelling catheter for the purpose of chemotherapy infusion No CNS metastases Hormone receptor status: Not specified

PATIENT CHARACTERISTICS: Age: 18 and over Sex: Female Menopausal status: Not specified Performance status: Karnofsky 70-100% Life expectancy: Not specified Hematopoietic: Hemoglobin at least 9.0 g/dL WBC at least 3,000/mm3 Platelet count at least 100,000/mm3 Granulocyte count at least 1,500/mm3 Hepatic: Bilirubin no greater than 1.5 times upper limit of normal (ULN) ALT, AST, and alkaline phosphatase no greater than 2.5 times ULN (no greater than 4.0 times ULN with liver or bone metastases) Renal: Creatinine no greater than 1.5 times ULN Cardiovascular: No clinically significant cardiovascular disease (e.g., uncontrolled hypertension, myocardial infarction, unstable angina, intractable arrhythmia, congestive heart failure, or New York Heart Association class II-IV heart disease) Left ventricular ejection fraction at least 50% or above lower limit of normal, whichever is lower Other: No severe hypersensitivity to products containing Cremophor EL (e.g., cyclosporine or teniposide for injection concentrate) No other serious medical condition that would preclude study Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 14 days since prior immunotherapy No prior trastuzumab (Herceptin) No other concurrent immunotherapy Chemotherapy: See Disease Characteristics Prior cytotoxic chemotherapy allowed in adjuvant setting Prior cumulative doxorubicin exposure no greater than 300 mg/m2 At least 1 year since prior taxane therapy No other concurrent chemotherapy Endocrine therapy: At least 14 days since prior hormonal therapy No concurrent hormonal therapy (e.g., tamoxifen, megestrol acetate, fluoxymesterone, or aminoglutethimide) Radiotherapy: At least 14 days since prior radiotherapy No concurrent radiotherapy to target lesions Surgery: Not specified Other: At least 30 days since other prior investigational agent or procedure No other concurrent investigational agents

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-01; Primary Completion 2001-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew D. Seidman, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States